CLINICAL TRIAL: NCT04945382
Title: Evaluation of the Retention of a Flowable Resin-based Sealant With Two Types of Adhesives in First Permanent Molars. A Randomized Clinical Trial in 12 Months
Brief Title: Retention of a Flowable Resin-based Sealant With Two Types of Adhesives
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University of San Marcos, Peru (Other)
Responsible Party: Principal Investigator, Gilmer Torres Ramos, DDS,PhD, National University of San Marcos, Peru
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: A20052171
Record Dates: First submitted 2021-06-15; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Caries,Dental; Pit and Fissure Caries; Sealant Dental
MeSH Terms: conditions — Dental Caries; Van der Woude syndrome

STUDY DESIGN:
Intervention Model Description: A split mouth study design will be adopted , which consists of a simple division of the mouth into two parts (right and left) for the first four permanent molars of each patient, where the placement of the materials will be on the right / left side of the mouth and contralateral. They will then be randomly assigned following block randomization procedures with a 1: 1 allocation using the random block sizes of 4 and 8. A computerized random number generator and combinations will be used to select the tooth and material to be sealed first.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scotchbond universal 3M (Experimental): Application of dental sealant with Scotchbond universal 3M adhesive.
  Interventions: Device: Scotchbond Universal 3M
- Control (Single bond 3M) (Active Comparator): Application of dental sealant with Single Bond 3M adhesive
  Interventions: Device: Single Bond 3M

INTERVENTIONS:
Device: Scotchbond Universal 3M — The occlusal surfaces will be cleaned using water, a brush and a low-pressure handpiece; they will wash and dry; then deproteinization will be done with sodium hypochlorite (5.25%) for 60 seconds, it will be washed with a water / air spray for 30s; it will dry up; The tooth will then be etched using a 37% orthophosphoric acid gel for 15 seconds, rinsed with a water / air spray for 30 seconds, and dried with cotton balls. Scotchbond universal 3M to the etched surface will be dried under a gentle air flow for 2-3 s, and light cured for 11 s using an LED curing unit with an output of 1500 mW / cm2 (Balloon.).
  Arms: Scotchbond universal 3M
Device: Single Bond 3M — The occlusal surfaces will be cleaned using water, a brush and a low-pressure handpiece; they will wash and dry; then deproteinization will be done with sodium hypochlorite (5.25%) for 60 seconds, it will be washed with a water / air spray for 30s; it will dry up; The tooth will then be etched using a 37% orthophosphoric acid gel for 15 seconds, rinsed with a water / air spray for 30 seconds, and dried with cotton balls. Single Bond 3M to the etched surface will be dried under a gentle air flow for 2-3 s, and light cured for 11 s using an LED curing unit with an output of 1500 mW / cm2 (Balloon.).
  Arms: Control (Single bond 3M)

SUMMARY:
The aim of the present study is to compare the use of two adhesives for the placement of occlusal sealants, evaluating their retention on the occlusal surfaces. Methods: A randomized clinical trial, in Phase IV, triple-blind, with a split mouth study design will be adopted, which consists of a simple division of the mouth into two parts (right and left) for the first four permanent molars of each patient, where the placement of the materials will be on the right / left side of the mouth and contralateral. They will then be randomly assigned following block randomization procedures with a 1: 1 allocation. 50 participants (6-year-old children) will be considered, and a pair of permanent first molars homologs will be used for each participant. Inclusion criteria include: children whose parents accepted their participation in the study and who signed the Informed Consent, children enrolled in the Pichanaki District school, children who present upper and / or lower permanent molars with absence of deep caries cavities and caries, graded 0 and 1 according to ICDAS II, Green and Vermillion Simplified Oral Hygiene Index of 1-2, have a pair of non-cavitated caries-free counterparts, and children with positive behavior. After selection of patients, the dental sealants will be placed with two different adhesives: the 8th generation adhesive intervention group (Scotchbond universal 3M) and the 5th generation adhesive control group (Single bond 3M), both sealants will use the same flowable resin (Tetric N-flow ivoclar vivadent). Results evaluation: Retention of the sealants will be evaluated at 6, 9 and 12 months. Retention rates of pit and fissure sealant materials will be analyzed according to the split mouth design. The study will use the Mc Nemar test to compare the retention of sealants in the intervention group and the control group at 6, 9 and 12 months. A 95% confidence level will be accepted. In addition, the Cochrane Q test will be applied to determine if there are significant differences in survival for each group of sealants through the evaluation time. The calculation of the survival months of the sealants will be carried out using the actuarial method (survival tables). Expected conclusion: To identify which of the two adhesives presents the best retention after 12 months.

DETAILED DESCRIPTION:
Ethical considerations This research will be carried out in a Pichanaki District school, at Chanchamayo province, for which we will request the review by the Research Ethics Committee of the Institute of Tropical Medicine "Daniel Alcides Carrión" UNMSM, in addition to process the permits to the pertinent authorities of the school of the Pichanaki province (verbal and written) on the principles of the treatment, the risks of the procedures and the purpose of the study, and the parents or guardians of the participants will sign the consent forms informed appropriate. Type and Research Design A split mouth study design will be adopted, which consists of a simple division of the mouth into two parts (right and left) for the first four permanent molars of each patient, where the placement of the materials will be on the right / left side of the mouth and contralateral. Study population 6-year-olds from kindergarden 380 of Pichanaqui, Junin department Sample size 50 participants. A pair of permanent first molars homologs will be used for each participant.Data collection techniques Coordination with the Ethics and Parental Authorization Committee Letters of invitation will be made and they will be distributed in class through the teachers, and each student will take it home to deliver to their parents or guardians. Each letter (envelope) will have the informed consent, the informed assent, data record sheet and an informative bulletin where it explains all the procedure that will be carried out for each participant, there will also be an informative talk in the school for parents and teachers, where they will be informed about the study and will collect the envelopes. The research team will not force any child to participate; each will have the option to choose to participate in the study by verbal assent. A report will be delivered to the parent or guardian of the child after the intervention. Recruitment of participants Participants will be recruited within the month the invitation letters will be delivered. Informed consent process Researcher 1 will give an informative talk about the study and will collect the envelopes containing the informed consent, informed consent and data record sheet). Students and parents who accept participation will receive a summons for subsequent dental visits. It will collect the consents signed by both parents / guardians and in case the signature of one of the parents cannot be obtained either due to impossibility (Death, difficulty in obtaining the signature, absence and reasons of personal strength). Only the signature of one will be accepted to give consent; and informed assent if the child reports that he understands and is mature enough to understand. Diagnostic Process Assistant 1 will be in charge of bringing the students for their dental check-up and will also provide the materials to operator 1 who will do the oral hygiene and prophylaxis index procedure. Afterwards, operator 2 will be previously calibrated according to the ICDAS II criteria, using the visual method it will detect and classify the lesions according to the International System criteria. Detection and Evaluation of Caries (ICDAS-II) and the teeth that will represent scores 0 and 1 will be selected. The inclusion and exclusion criteria mentioned above will be taken into account; and patients who have at least one pair of homologous permanent first molars that meet the same requirements will be considered. The maid 2 will be in charge of filling out the data sheets of the participants. Operator 1 will evaluate the Simplified Oral Hygiene Index until you reach an OHI score of 1-2 over a period of one month. Researcher 1 will select the participants taking into account the inclusion and exclusion criteria and will deliver the list of those participants to the programmer for randomization. Randomization Process There will be a programmer without participation in the clinical trial who will do the randomization sequence, will generate a list of numbers randomly assigned to participants and will be created with Stata 16 statistical software (Stata Corp. College Station, TX). The sample will be stratified by gender. They will then be randomly assigned following block randomization procedures. with a 1: 1 allocation using the random block sizes of 4 and 8, a computerized random number generator and combinations will be used to select the tooth and material to be sealed first. The Adhesive will be placed in a dispenser and will be coded by letters (A and B) the 8th generation adhesive intervention group (Scotchbond universal 3M) and the 5th generation adhesive control group (Single bond 3M), both sealants will use the same fluid resin (Tetric N-flow ivoclar vivadent). The name of each participant will be coded by numbers, this will be done by the programmer; the materials are going to be encoded letters (A and B) and the cards are going to be worked with these encodings for later data analysis.And with respect to the patient's data, it will only be handled by the programmer who will be in charge of coding, randomizing the first permanent molars, randomizing the materials to be used so that it is placed in the first permanent molars and this information will be given to the coordinator so that the put in sealed envelopes and then these sealed envelopes will be given to an assistant so that such data is not disclosed or published. In case this section of data confidentiality is in the informed consent it could be mentioned. The programmer will give the randomized list to the coordinator and the coordinator will give the external assistant not participating in the clinical trial in sealed envelopes labeled by each participant. This external assistant will take the randomized patient for treatment. Allocation concealment mechanism process and implementation The programmer will give this list generated to the coordinator and an external assistant will receive the envelopes with the same characteristics and will be in charge of taking the patient to receive treatment. Blinding process Blinding and balancing will be strictly maintained; by emphasizing the operators, assistants, evaluators, workers of the educational institution and the parents / guardians and participants. While the participants, operators, evaluators, assistants assigned to carry out the diagnosis, procedure and placement of the material, will not know the brand of the adhesives for pits and fissures, due to that they will be in a dispenser with code (A and B). Outcome assessors and data analysts will be blinded to allocation. Investigators who performed the intervention procedure will not take the results measures. Procedures process The external assistant to the study will be in charge of placing in the dispenser and listing the intervention material A (Scotchbond universal 3M) and B (single bond 3M) in prior coordination with the research coordinator. Operator 3 and assistant 4 will be previously trained and calibrated; they will do the procedure, without knowing the names of the stickers. Devices will be applied in the upper / lower first molars with adhesive, being the order assigned according to the previous randomization, for the intervention group they will be sealed by applying 8th generation adhesive (Scotchbond universal 3M) with a fluid resin (Tetric N-Flow) and on the contralateral side the upper / lower first molars will be sealed, the control group will be applied with a fifth generation adhesive (3M single bond) with a fluid resin (Tetric N-Flow ) Placement of materials on the right / left side of the mouth will be randomly assigned. A total of 100 upper / lower molar teeth will be sealed with both materials (50 teeth for each material). The materials will be placed by the same operator according to the protocol of Dr. Gilmer Torres Ramos for sealing pits and deep fissures. Steps for the application of the sealant, the teeth will be isolated with cotton rolls carefully and the assistant 4 will hold a plastic saliva ejector to avoid contamination of the saliva and facilitate the operative procedures of the occlusal surfaces of the upper molars and / or lower for each operator: The occlusal surfaces will be cleaned using water, a brush and a low-pressure handpiece; they will wash and dry; then deproteinization will be done with sodium hypochlorite (5.25%) for 60 seconds, it will be washed with a water / air spray for 30s; it will dry up; The tooth will then be etched using a 37% orthophosphoric acid gel for 15 seconds, rinsed with a water / air spray for 30 seconds, and dried with cotton balls. universal 3M) to the etched surface will be dried under a gentle air flow for 2-3 s, and light cured for 11 s using an LED curing unit with an output of 1500 mW / cm2 (Balloon.). and for the control group, a 5th generation adhesive (SINGLE BOND 3M) will be applied to the etched surface, it will be dried under a gentle air flow for 2-3 s, and it will be light-cured for 11 s using an LED curing unit. with an output of 1500 mW / cm2 (Balloon.), then a uniform layer will be applied to both groups, a sealant based on fluid resin (Tetric N-Flow ivoclar vivadent) will be light-cured for 11 s using an LED curing unit with an output 1500 mW / cm2 (Balloon). The cotton rolls and plastic saliva ejector will be removed, and the occlusion will be checked with articulating paper. The operator will not know the brand of adhesive to be used, because it will be in the dispenser and will be delivered by another person (external assistant to the study) previously trained for this activity and both materials have a similar color. The child will also not be informed about the brand of the material used. The assistant 5 will collect the data on the card. An average attendance will be 6 participants per day with time intervals to prepare the work environment between each procedure. Evaluation and monitoring process Assistant 6 will bring and take the participants to operator 4 who will do the prophylaxis and help fill out the cards. Operator 5 with at least ten years of experience will be previously trained, evaluated and calibrated; in accordance with ICDASS II criteria and retention of sealants. The calibration will be given by the Kappa measure (κ > 0.7). Operator 5 will not have performed the pit and fissure sealants procedure; he will record the retention of the sealant in a period of 6, 9 and 12 months. Followup of sealed teeth will be observed with good lighting, after tooth prophylaxis. It will be evaluated with an oral mirror and periodontal probe. Each sealant is classified as Total retention of the sealant in all pits and fissures (TR); Partial retention of the sealant in some pits and fissures (PR); Total loss of sealant in all pits and fissures (TL) The coordinator will be in all evaluation follow-ups. Analysis and interpretation of information A descriptive analysis of the study population will be made, where the qualitative variables will be represented with absolute frequencies and percentages. With the registration cards a database will be built (Excel software Version 18.0), retention rates of pit and fissure sealant materials will be analyzed using SPSS software 23. An analysis will be performed according to the split mouth design. This design proposes two types of analysis as qualitative or binary measure. For the binary modality, the Mac Nemar Chi-square test is recommended. The study will use the Mc Nemar test to compare the retention of sealants in the intervention group and the control group used at 6, 9 and 12 months. A 95% confidence level will be accepted. In addition, the Cochrane Q test will be applied to determine if there are significant differences in survival for each group of sealants through the evaluation time (6, 9 and 12 months). The calculation of the survival months of the sealants will be carried out using the actuarial method (survival tables)

ELIGIBILITY:
Inclusion Criteria:

* Children whose parents accepted their participation in the study and who signed the Informed Consent
* Children enrolled in the Pichanaki District school, Chanchamayo province, in Junin department 6-year-old children, who present upper and / or lower permanent molars with the following characteristics:

  * Absence of deep caries cavities and caries, graded 0 and 1 according to ICDAS II
  * Green and Vermillion Simplified Oral Hygiene Index (OHI) of 1-2
  * Have a pair of non-cavitated caries-free counterparts.
* Children with positive behavior.

Exclusion Criteria:

* Children with the presence of a deep dental caries lesion, with pulp exposure, history of pain and presence of fistula or abscess adjacent to decayed tooth. • Medically compromised children
* Children with developmental enamel defects.
* Children with a known allergy to any of the resins used
* Children with previously placed sealants or restorations
* Children residing outside the city

Ages: 72 Months to 83 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Clinical Retention of adhesives | 12 months
  Determine which of the two adhesives has better clinical retention during the period of 12 months, one with Scotchbond Universal 3M adhesive and the other with Single bond 3M adhesive.

SECONDARY OUTCOMES:
Clinical preservation of sealats | 12 months
  Evaluate the clinical preservation of one sealant with Scotchbond Universal 3M adhesive and another sealant with Single Bond 3M adhesive, in first permanent molars, in the period of 12 months.
.Survival curve of sealants | 12 months
  Estimate the survival curve of one sealant with Scotchbond Universal 3M adhesive and another sealant with Single Bond 3M adhesive, in first permanent molars, in the period of 12 months.
Survivability of sealant | 12 months
  Compare the survivability of a sealant with Scotchbond Universal 3M adhesive and another sealant with Single Bond 3M adhesive, in first permanent molars, in the period of 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Nido 380, Alto Pichanaki, Chanchamayo, Peru

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Alirezaei M, Bagherian A, Sarraf Shirazi A. Glass ionomer cements as fissure sealing materials: yes or no?: A systematic review and meta-analysis. J Am Dent Assoc. 2018 Jul;149(7):640-649.e9. doi: 10.1016/j.adaj.2018.02.001. Epub 2018 May 4. PMID 29735163
- [Result] Aman N, Khan FR, Salim A, Farid H. A randomized control clinical trial of fissure sealant retention: Self etch adhesive versus total etch adhesive. J Conserv Dent. 2015 Jan-Feb;18(1):20-4. doi: 10.4103/0972-0707.148883. PMID 25657521
- [Result] Dikmen B. Icdas II criteria (international caries detection and assessment system). J Istanb Univ Fac Dent. 2015 Oct 21;49(3):63-72. doi: 10.17096/jiufd.38691. eCollection 2015. PMID 28955548
- [Result] Ekstrand KR, Gimenez T, Ferreira FR, Mendes FM, Braga MM. The International Caries Detection and Assessment System - ICDAS: A Systematic Review. Caries Res. 2018;52(5):406-419. doi: 10.1159/000486429. Epub 2018 Mar 8. PMID 29518788
- [Result] Gugnani N, Pandit IK, Srivastava N, Gupta M, Sharma M. International Caries Detection and Assessment System (ICDAS): A New Concept. Int J Clin Pediatr Dent. 2011 May-Aug;4(2):93-100. doi: 10.5005/jp-journals-10005-1089. Epub 2010 Apr 15. PMID 27672245
- [Result] Hou J, Gu Y, Zhu L, Hu Y, Sun M, Xue H. Systemic review of the prevention of pit and fissure caries of permanent molars by resin sealants in children in China. J Investig Clin Dent. 2017 Feb;8(1). doi: 10.1111/jicd.12183. Epub 2015 Aug 14. PMID 26272130
- [Result] Jafarzadeh M, Malekafzali B, Tadayon N, Fallahi S. Retention of a Flowable Composite Resin in Comparison to a Conventional Resin-Based Sealant: One-year Follow-up. J Dent (Tehran). 2010 Winter;7(1):1-5. Epub 2010 Mar 31. PMID 21998768
- [Result] Karaman E, Yazici AR, Tuncer D, Firat E, Unluer S, Baseren M. A 48-month clinical evaluation of fissure sealants placed with different adhesive systems. Oper Dent. 2013 Jul-Aug;38(4):369-75. doi: 10.2341/12-181-C. Epub 2012 Dec 4. PMID 23210859
- [Result] Khare M, Suprabha BS, Shenoy R, Rao A. Evaluation of pit-and-fissure sealants placed with four different bonding protocols: a randomized clinical trial. Int J Paediatr Dent. 2017 Nov;27(6):444-453. doi: 10.1111/ipd.12281. Epub 2016 Dec 26. PMID 28024165
- [Result] Maher MM, Elkashlan HI, El-Housseiny AA. Effectiveness of a self-etching adhesive on sealant retention in primary teeth. Pediatr Dent. 2013 Jul-Aug;35(4):351-4. PMID 23930635
- [Result] Rishika, Garg N, Mayall SS, Pathivada L, Yeluri R. Combined Effect of Enamel Deproteinization and Intermediate Bonding in the Retention of Pit and Fissure Sealants in Children: A Randomized Clinical Trial. J Clin Pediatr Dent. 2018;42(6):427-433. doi: 10.17796/1053-4625-42.6.4. Epub 2018 Aug 7. PMID 30085876
- [Result] Muller-Bolla M, Courson F, Lupi-Pegurier L, Tardieu C, Mohit S, Staccini P, Velly AM. Effectiveness of Resin-Based Sealants with and without Fluoride Placed in a High Caries Risk Population: Multicentric 2-Year Randomized Clinical Trial. Caries Res. 2018;52(4):312-322. doi: 10.1159/000486426. Epub 2018 Mar 1. PMID 29495020
- [Result] Fracasso Mde L, Rios D, Machado MA, Silva SM, Abdo RC. Avaliacao da microinfiltracao marginal e profundidade de penetracao dos cimentos de ionomero de vidro utilizados como selantes oclusais. J Appl Oral Sci. 2005 Sep;13(3):269-74. doi: 10.1590/s1678-77572005000300013. PMID 20878029
- [Result] Wadhwa S, A Nayak U, Kappadi D, Prajapati D, Sharma R, Pawar A. Comparative Clinical Evaluation of Resin-based Pit and Fissure Sealant and Self-adhering Flowable Composite: An In Vivo Study. Int J Clin Pediatr Dent. 2018 Sep-Oct;11(5):430-434. doi: 10.5005/jp-journals-10005-1552. Epub 2018 Oct 1. PMID 30787558
- [Result] Tandon V, Lingesha RT, Tangade PS, Tirth A, Pal SK, Lingesha CT, Arora V, Yadav V. Effect of Adhesive Application on Sealant Success: A Clinical Study of Fifth and Seventh Generation Adhesive Systems. J Dent (Tehran). 2015 Oct;12(10):712-9. PMID 27252754
- [Result] Topal BG, Kirzioglu Z. Evaluation of the fissure sealants applied to erupting permanent molars in accordance to eruption stages: A prospective study. Niger J Clin Pract. 2019 Nov;22(11):1495-1502. doi: 10.4103/njcp.njcp_534_18. PMID 31719270